CLINICAL TRIAL: NCT01752348
Title: Effects of Free Fatty Acids and 3-hydroxybutyrate on Protein, Glucose, Lipid Metabolism and Intracellular Signals; a Study on Muscle Wasting and Metabolism During Acute Inflammation and Potential Anabolic Mechanisms.
Brief Title: Effects of Free Fatty Acids and 3-hydroxybutyrate on Protein, Glucose, Lipid Metabolism and Intracellular Signals.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 11422796; 1-10-72-530-12 (Other: Regional Ethics Comite)
Record Dates: First submitted 2012-12-14; First posted 2012-12-19 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2013-07

CONDITIONS: Systemic Inflammatory Response Syndrome
Keywords: sepsis; cytokine release; fever
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Sepsis; Fever | interventions — Endotoxins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (isotonic saline) (Placebo Comparator): Endotoxin + isotonic saline. Reference for model of acute inflammatory illness
  Interventions: Other: Endotoxin, US standard reference E.coli
- Acipimox + Placebo (isotonic saline) (Experimental): Endotoxin + Acipimox + Placebo (isotonic saline). Intervention: blockage of endogenous lipolysis.
  Interventions: Other: Endotoxin, US standard reference E.coli
- Acipimox + free fatty acids (Experimental): Endotoxin + Acipimox + free fatty acids. Intervention: free fatty acids
  Interventions: Other: Endotoxin, US standard reference E.coli
- Acipimox + 3-hydroxybutyrate (Experimental): Endotoxin + Acipimox + 3-hydroxybutyrate. Intervention: 3-hydroxybutyrate
  Interventions: Other: Endotoxin, US standard reference E.coli

INTERVENTIONS:
Other: Endotoxin, US standard reference E.coli

SUMMARY:
The investigators hypothesize that the investigators can detect protein-sparing effects of administration of the ketone 3-hydroxybutyrate and free fatty acids during simulation of an acute inflammatory disease. The investigators use the infusion of endotoxin, US standard reference E.coli in healthy subjects as a model for inflammation / infection and to evaluate the effect on protein metabolism using different tracers and the investigators can measure the various intracellular signaling pathways of selected muscle and adipose tissue.

ELIGIBILITY:
Inclusion Criteria:

* 20 < body mass index < 30 kg/m2.
* written and orally informed consent before enrollment.

Exclusion Criteria:

* participation in other studies using radioactive tracers or other exposure to radiation (X-rays, scintigraphy etc).
* allergy to soy products or eggs
* diabetes, any type
* epilepsy
* ongoing infection
* immune deficiency
* cardiovascular disease
* dysregulated hypertension
* primary muscles disease, congenital or acquired

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2013-02; Primary Completion 2014-07 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Protein metabolism | 6 hours intervention period
  Measurements of protein oxidation during intervention using radioactive tracer techniques.

SECONDARY OUTCOMES:
Activated intracellular signalling pathways | study day
  Measurements on biopsies from muscle and fatty tissue taken on day of study

OTHER OUTCOMES:
Other systemic metabolic effects | 6 hours of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Niels Møller, Professor, Principal Investigator — Institute of Clinical Medicine, Aarhus University, Denmark. Department of Internal Medicin and Endocrinology, Aarhus university hospital, Aarhus, Denmark.
Locations (1):
- Medical Research Laboratory, Department of Internal Medicine and Endocrinology, Aarhus C, Denmark

REFERENCES:
- [Derived] Thomsen HH, Rittig N, Johannsen M, Moller AB, Jorgensen JO, Jessen N, Moller N. Effects of 3-hydroxybutyrate and free fatty acids on muscle protein kinetics and signaling during LPS-induced inflammation in humans: anticatabolic impact of ketone bodies. Am J Clin Nutr. 2018 Oct 1;108(4):857-867. doi: 10.1093/ajcn/nqy170. PMID 30239561